CLINICAL TRIAL: NCT02998229
Title: Artisse™ Intrasaccular Device IDE
Brief Title: The Artisse™ Intrasaccular Device is Indicated for the Treatment of Wide-neck Bifurcating Intracranial Aneurysms (IAs).
Acronym: ARTISSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT24004
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm; Intrasaccular; Artisse
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artisse™ Intrasaccular Device (Experimental): Study subjects with an unruptured or ruptured wide-neck bifurcating intracranial aneurysm will be treated by endovascular implantation of the Artisse™ Intrasaccular Device.
  Interventions: Device: Artisse™ Intrasaccular Device

INTERVENTIONS:
Device: Artisse™ Intrasaccular Device — Intrasaccular Device

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Artisse™ Intrasaccular Device in the treatment of unruptured and ruptured wide-neck bifurcating intracranial aneurysms.

DETAILED DESCRIPTION:
The Artisse™ IDE study is a prospective, multi-center, single-arm Investigational Device Exemption (IDE) study of the Artisse™ Intrasaccular Device for the treatment of IAs. The primary objective of the Artisse™ IDE study is to assess the safety and effectiveness of the Artisse™ Intrasaccular Device in the treatment of unruptured and ruptured wide-neck bifurcating intracranial aneurysms. The effectiveness of the Artisse™ Intrasaccular Device is measured by its ability to completely occlude the treated aneurysm without retreatment of the target aneurysm, recurrent subarachnoid hemorrhage from the target aneurysm, or significant parent artery stenosis (> 50% stenosis) at 1 year post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's Legally Authorized Representative (LAR) has provided written informed consent using the Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent Form (ICF). Health Insurance Portability and Accountability Act (HIPAA)/data protection authorization has been provided and signed by the subject or subject's LAR.
2. Subject is 18-75 years of age at the time of consent.
3. Subject has a single unruptured or ruptured IA requiring treatment. If the patient has an additional IA, the additional IA must not be deemed to require treatment within 1-year of the index procedure.
4. The target aneurysm must have the following characteristics:

   1. Saccular morphology
   2. Located at a bifurcation in the anterior or posterior circulation
   3. Aneurysm Width appropriate for treatment with the Artisse™ Intrasaccular Device for device sizingper the Instructions for Use.
   4. Wide-necked, defined as neck size ≥ 4 mm and/or a dome-to-neck ratio of ≥ 1 and < 2.
5. If the target aneurysm was acutely ruptured, subject must be neurologically stable with Hunt and Hess Grade of I or II.

   Ruptured IA is defined as showing evidence of SAH attributed to the target aneurysm within the last 30-days (using computed tomography (CT), magnetic resonance imaging (MRI), or lumbar puncture (LP).)
6. Subject is able to comply with all aspects of the Clinical Investigation Plan (CIP) requirements (e.g., screening, evaluation, treatment, and the post-procedure follow-up schedule).
7. Subject meets one or more risk factors for IA rupture, such as age, hypertension, cigarette smoking, use of sympathomimetic drugs, Japanese or Finnish ancestry, history of prior aneurysmal subarachnoid hemorrhage (aSAH), familial intracranial aneurysms or SAH, clinical or radiological mass effect, reduced quality of life due to fear of rupture, IA size, location, and morphology, documented growth of IA on serial imaging (or enhanced aneurysm walls on contrast), presence of multiple IAs, and presence of concurrent pathology.
8. Treating physician has already selected the subject for endovascular treatment of the target aneurysm after considering risk-benefit of clipping vs endovascular treatment
9. If the subject has an additional IA that was treated previously, the additional IA must have been clinically stable in the past 90 days (i.e. without ongoing adverse events related to the previous treatment).

Exclusion Criteria:

1. During treatment planning, it is determined that subject may need an adjunctive implant device in addition to the Artisse™ Intrasaccular Device. (Subjects who need unplanned adjunctive implant devices are not excluded.)
2. Subject's target aneurysm was previously treated with other devices/implants (e.g., coils) or parent artery has a stent or other obstruction that could interfere with the correct placement of the Artisse™ Intrasaccular Device.
3. Subject has a known active systemic bacterial infection.
4. Subject has anatomy or physiology considered unsuitable (e.g., vessel anomaly or disease) for endovascular treatment with the Artisse™ Intrasaccular Device by the treating physician.
5. Subject has a mRS score > 2 (i.e., mRS scores of 3 to 5) prior to procedure (in case of unruptured IA) or prior to rupture (in case of ruptured IA).
6. Subject has an SAH from a non-target aneurysm or any other intracranial hemorrhage within 90 days.
7. Subject, of child-bearing potential, is pregnant (confirmed with a positive pregnancy test) or plans to become pregnant during the 1 year follow up period after the index procedure.
8. Subject is enrolled in another device or drug study in which participation could confound study results.
9. The treating physician determines that the health of the subject or the validity of the study outcomes (e.g., high risk of neurologic events, conditions that may increase the chance of stroke) may be compromised by the subject's enrollment.
10. Subject has a known hypersensitivity, which cannot be medically treated, to any component of the study device, procedural materials, or medications commonly used during the procedure.
11. Subject is taking anticoagulants (e.g., warfarin) that cannot be discontinued for a minimum of 7 days post-procedure or have a known blood dyscrasia, coagulopathy, or hemoglobinopathy.
12. Subject has acute or chronic renal failure (unless on dialysis) that would prevent them from undergoing digital subtraction angiography (DSA).
13. Subject has a life expectancy of less than 5 years due to an illness or condition other than the index IA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Incidence of complete aneurysm occlusion | 1 year post procedure
  Incidence of complete aneurysm occlusion without retreatment of the target aneurysm, recurrent subarachnoid hemorrhage (SAH) from the target aneurysm, or significant parent artery stenosis (>50% stenosis) at 1 year post-procedure.
Safety Evaluation | through study completion, an average of 5 years
  The safety of the Artisse™ Intrasaccular Device will be determined based on a review of all the serious adverse events (SAEs) observed during the study.

SECONDARY OUTCOMES:
Incidence of implant success | Procedure
  Proportion of subjects with device implant success at the target site
Incidence of recurrence | 1 year post procedure
  Proportion of subjects with angiographic aneurysmal recurrence at 1 year post-procedure
Incidence of stroke | 30 days, 180 days, 1 year, 3 years, and 5 years post-procedure
  Proportion of subjects experiencing a stroke (ischemic or hemorrhagic) within 30 days post-procedure, 180 days post-procedure, 1 year post-procedure, 3 years post-procedure, and 5 years post-procedure
Change in Modified Rankin Score (mRS) compared to baseline. mRS scores can range from 0 (no symptoms) to 5 (severe disability) with a separate category of 6 added for patients who expire. | 30 days, 180 days, 1 year, 3 years, and 5 years post-procedure
  Proportion of subjects with unruptured intracranial aneurysms (IAs) experiencing improvement, deterioration, or no change in the mRS score compared to baseline through 30 days post-procedure, 180 days post procedure, 1 year post-procedure, 3 years post-procedure, and 5 years post-procedure
Incidence of good clinical outcomes in unruptured intracranial aneurysms (IAs) | 30 days, 180 days, 1 year, 3 years, and 5 years post-procedure
  Proportion of subjects with unruptured IAs experiencing good clinical outcomes, defined as an Modified Rankin Score (mRS) score of 0-2 (0: No symptoms, 1: No significant disability despite symptoms, 3: Slight disability) through 30 days post-procedure, 180 days post-procedure, 1 year post-procedure, 3 years post-procedure, and 5 years post-procedure
Incidence of good clinical outcomes in ruptured intracranial aneurysms (IAs) | 30 days, 180 days, 1 year, 3 years, and 5 years post-procedure
  Proportion of subjects with ruptured IAs experiencing good clinical outcomes, defined as an Modified Rankin Score (mRS) score of 0-2 (0: No symptoms, 1: No significant disability despite symptoms, 3: Slight disability) through 30 days post-procedure, 180 days post-procedure, 1 year post-procedure, 3 years post-procedure, and 5 years post-procedure
Incidence of adequate aneurysm occlusion | 180 days, 1 year, 3 years, and 5 years post-procedure
  Incidence of adequate aneurysm occlusion of the target aneurysm at 180 days post-procedure, 1 year post-procedure, 3 years post-procedure, and 5 years post-procedure
Incidence of retreatment | 3 years and 5 years post-procedure
  Incidence of retreatment of the target aneurysm through 3 years post-procedure, and 5 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Harsh Sancheti, Study Director — Medtronic
Locations (18):
- United States (18):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albany Medical Center, Albany, New York
  - Buffalo General Medical Center, Buffalo, New York
  - The Mount Sinai Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Novant Health Brain and Spine Surgery, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Semmes Murphy Clinic, Memphis, Tennessee
  - University of Utah Hospital, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No